CLINICAL TRIAL: NCT02747628
Title: Comparative Study Between Transdermal Nicotine and Melatonin Patches on Postoperative Pain Relief After Laparoscopic Cholecystectomy, a Double-blind, Placebo-controlled Trial
Brief Title: Transdermal Nicotine and Melatonin Patches for Postoperative Pain Relief
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Dr., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 942
Record Dates: First submitted 2016-04-01; First posted 2016-04-22 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Pain Relief
Keywords: Transdermal nicotine; Transdermal melatonin; Postoperative pain; Laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- C group, (n=20) (Placebo Comparator): C group (n=20) (placebo group) each patient received transdermal placebo patch, identical placebo patches custom-made by 1-800-Patches (Salt Lake City, UT) placed 2 hours preoperatively for acute postoperative pain after laparoscopic cholecystectomy.
  Interventions: Drug: Placebo
- TDN group, (n=20) (Active Comparator): TDN group (n=20) each patient received transdermal therapeutic system- nicotine (15 mg/16 h),Nicorette® invisi 15mg patch releasing 15mg of nicotine over 16h, produced by Lohmann Therapie-System, Germany placed 2 hours preoperatively for acute postoperative pain after laparoscopic cholecystectomy.
  Interventions: Drug: transdermal therapeutic system- nicotine.
- TDM group, (n=20) (Active Comparator): TDM group (n=20) each patient received transdermal therapeutic system- melatonin (7 mg/8h),melatonin sleep patch from Respro Labs ™ containing 7 mg of melatonin placed 2 hours preoperatively for acute postoperative pain after laparoscopic cholecystectomy.
  Interventions: Drug: transdermal therapeutic system- melatonin.

INTERVENTIONS:
Drug: Placebo — Postoperative pain was evaluated based on visual analogue scale, first time to ask for rescue analgesia and total pethidine requirements (mg) in 12 hours postoperatively were also recorded.
  Arms: C group, (n=20)
Drug: transdermal therapeutic system- nicotine. — Postoperative pain was evaluated based on visual analogue scale, first time to ask for rescue analgesia and total pethidine requirements (mg) in 12 hours postoperatively were also recorded.
  Other Names: TDN, Nicorette® invisi 15mg /16hr.
  Arms: TDN group, (n=20)
Drug: transdermal therapeutic system- melatonin. — Postoperative pain was evaluated based on visual analogue scale, first time to ask for rescue analgesia and total pethidine requirements (mg) in 12 hours postoperatively were also recorded.
  Other Names: TDM, melatonin sleep patch from Respro Labs ™ (7 mg/8hr).
  Arms: TDM group, (n=20)

SUMMARY:
Sixty female non-smoker patients, aged 18-50 years and ASA I and II undergoing elective laparoscopic cholecystectomy under general anesthesia were included in this randomized controlled double-blind study. Patients were randomly divided into 3 groups 20 each, C group patients received transdermal placebo patch, TDN group (15 mg/16 h) and TDM group (7 mg/8h). Assessment of postoperative pain, sedation, hemodynamic variables such as HR and MAP, postoperative monitoring of arterial SpO2 and side effects (e.g. nausea, vomiting, pruritis, respiratory depression and hemodynamic instability) were done 30 minutes, 1, 2, 6 and 12 hours postoperatively. Postoperative Patient's and Surgeons' satisfaction, Intraoperative bleeding and plasma cortisol (µg / dl) 2 hours postoperatively were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* 60 female patients.
* non-smoker patients.
* aged between 18 and 50 years old.
* ASA physical status I and II.
* 70-90 kg body weight and height 160-180 cm.
* undergoing elective laparoscopic cholecystectomy under general anesthesia.

Exclusion Criteria:

* Patients with impaired kidney or liver functions.
* history of cardiac or central nervous system disease.
* history of smoking.
* history of drug or alcohol abuse.
* history of chronic pain or daily intake of analgesics.
* uncontrolled medical disease (diabetes mellitus and hypertension).
* history of intake of non-steroidal anti-inflammatory drugs or opioids within 24 h before surgery.
* allergy to the used medications.
* coagulation defect.
* local infection at the site of application of transdermal patch.
* patient's refusal.
* duration of surgery more than 120 minutes.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | C Group, (n=20) | TDN Group, (n=20) | TDM Group, (n=20)
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | C Group, (n=20) | TDN Group, (n=20) | TDM Group, (n=20) | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (3.39) | 43.1 (2.4) | 44.3 (1.86) | 43.2 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 20 | 60
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 20 | 20 | 20 | 60
Duration of anesthesia (min) [Mean (Standard Deviation); unit: minutes] | 111.2 (3.4) | 112.8 (4.4) | 111.4 (3.78) | 111.8 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: A Mean Difference of Total Analgesic (Pethidine) Consumption.
Time Frame: [Time Frame: The total pethidine requirements (mg) 12 hours postop]
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | C Group, (n=20) | TDN Group, (n=20) | TDM Group, (n=20)
Number analyzed (Participants) | 20 | 20 | 20
mg | 122.15 (6.38) | 55.5 (3.97) | 59.7 (4.43)

ADVERSE EVENTS:
Arm/Group | C Group, (n=20) | TDN Group, (n=20) | TDM Group, (n=20)
Serious Adverse Events (participants affected / at risk) | 0/20 | 4/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 8/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C Group, (n=20) (N=20) | TDN Group, (n=20) (N=20) | TDM Group, (n=20) (N=20)
Vomiting (Gastrointestinal disorders) | 0 | 4 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C Group, (n=20) (N=20) | TDN Group, (n=20) (N=20) | TDM Group, (n=20) (N=20)
nausea (Gastrointestinal disorders) | 0 | 8 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No